CLINICAL TRIAL: NCT03493607
Title: An Open-label Study to Investigate the Safety, Tolerability and Efficacy of a Single 6-hour Intravenous Infusion of AMO-01 to Treat Adolescents and Adults With Phelan-McDermid Syndrome (PMS) and Co-morbid Epilepsy
Brief Title: AMO-01 to Treat Adolescents and Adults With Phelan-McDermid Syndrome (PMS) and Co-morbid Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexander Kolevzon (Other)
Responsible Party: Sponsor-Investigator, Alexander Kolevzon, Clinical Director, Associate Professor, Seaver Autism Center for Research and Treatment, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-2226
Record Dates: First submitted 2018-04-04; First posted 2018-04-10 (Actual); Results first posted 2021-06-22 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Phelan-McDermid Syndrome; Epilepsy
Keywords: AMO-01; Shank3; Clinical Trial
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome; Epilepsy

STUDY DESIGN:
Intervention Model Description: Single Group, open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMO-01 (Experimental): Intravenous Infusion
  Interventions: Drug: AMO-01

INTERVENTIONS:
Drug: AMO-01 — Subjects will receive a single 6-hour intravenous infusion for a total dose administration or 120 mg/m2 of AMO-01.

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and efficacy of a single 6-hour intravenous infusion of AMO-01 to treat adolescents and adults with PMS and co-morbid epilepsy. Phelan-McDermid Syndrome (PMS) is a neurodevelopmental disorder characterized by a chromosomal deletion or mutation at 22q13.3 that contains the SHANK3/ProSAP2 gene. A key co-morbidity in PMS is the presence of epilepsy. Currently there are no approved treatments for PMS. Furthermore, there has been relatively little clinical study of pharmacological interventions for PMS. AMO-01 may provide benefit to PMS patients exhibiting behavioral abnormalities and seizures.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects under study must have a diagnosis of Phelan McDermid syndrome (PMS) with genetic confirmation of pathogenic SHANK3 deletion or mutation.
2. Subjects must be post pubertal males or females aged ≥12 years and ≤45 years at Screening.
3. Subject must have a diagnosis of epilepsy.
4. Subjects must have a syndrome-specific Clinical Global Impression- Severity Score of 4 or greater at Screening
5. Subject's parent or legally authorized representative (LAR) must provide written informed consent before any study related procedures are conducted. Where a parent or LAR provides consent, there must also be assent from the subject (as required by local regulations).
6. Subject's caregiver must be willing and able to support the subject's participation for the duration of the study.
7. Subject's caregiver is able and willing to maintain an accurate and complete daily written seizure diary for the entire duration of the study.

Exclusion Criteria:

1. Receiving medications/therapies not stable (i.e. changed) within 4 weeks prior to Screening. For each enrollee, every effort should be made to maintain stable regimens of allowed concomitant medications and allowed non -medicine based therapies throughout the course of the study, from Screening until the last study assessment.
2. Known hypersensitivity to farnesylated dibenzodiazepinone or any of the formulation components.
3. Subjects with a history of uncontrolled hypotension or hypertension (Polysorbate 80 is a major constituent of AMO-01 and can cause hypotension).
4. Subjects that have received Coumadin or heparin in the 2 weeks preceding Screening.
5. Medical illness or other concern which would cause the investigator to conclude that the subject will not be able to perform the study procedures or assessments or would confound interpretation of data obtained during assessments.
6. Females who are pregnant, lactating or not willing to use a protocol-defined acceptable contraception method if sexually active and not surgically sterile.
7. Males, engaged in sexual relations with a female of child bearing potential, not using an acceptable contraception method if sexually active and not surgically sterile.
8. Clinically significant abnormalities in safety laboratory tests, vital signs or ECG, as measured at Screening (may repeat to confirm).
9. Current clinically significant (as determined by the investigator) neurological, cardiovascular, renal, hepatic, endocrine or respiratory disease that may impact the interpretability of the study results.
10. Current clinically significant (as determined by the investigator) lymphedema that may compromise venous access and/or may have an adverse impact on study drug distribution and clearance.
11. Judged clinically to be at risk of suicide by the investigator.
12. Average QTcF value of >450 msec at Screening (may repeat to confirm).
13. Subjects in whom an indwelling intravenous line could not be established or maintained.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kolevzon, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Seaver Autism Center for Research and Treatment at Mount Sinai, New York, New York
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in Feb 2017, with first enrollment in May of 2018. Study was opened for enrollment through Jan 2021 when decision was made to close study due to low enrollment. Participants completed study visits. Last participant seen March 2020.
Groups:
- AMO-01: Subjects received a single 6-hour intravenous infusion for a total dose administration or 120 mg/m2 of AMO-01.
Period: Overall Study
Arm/Group | AMO-01
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AMO-01
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.6 (2.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: An adverse event is defined as any untoward medical occurrence in a study subject, temporally associated with the use of the experimental medication, whether or not considered related to the medication. An adverse event can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of the experimental medication. Adverse events will be monitored throughout all 8 weeks of study participation.
Time Frame: 8 weeks
Measure: Number; unit: events
Arm/Group | AMO-01
Number analyzed (Participants) | 6
events | 19

2. Secondary Outcome: Number of Weekly Seizure Counts
Description: Seizure frequency was measured by a caregiver-completed seizure diary throughout the duration of the trial. A seizure diary was provided to each family at the screening visit to record each seizure event, its date/time, duration, and type. The study team reviewed the diary at each visit with the caregiver and weekly seizure frequency was calculated.
  The week 1 seizure count was the number of seizures in the 7 days following the infusion day. Similarly, the week 2 seizure count was the number of seizures in the 7 days between weeks 1 and 2. Lastly, the week 4 seizure count was the sum of seizures in the 14 days between weeks 2 and 4, divided by 2.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: seizure event
Groups:
- Participants With Phelan-McDermid Syndrome (PMS) at Baseline: Participants with Phelan-McDermid syndrome (PMS) at baseline
- Participants With Phelan-McDermid Syndrome (PMS) at Week 1: Participants with Phelan-McDermid syndrome (PMS) at week 1
- Participants With Phelan-McDermid Syndrome (PMS) at Week 2: Participants with Phelan-McDermid syndrome (PMS) at week 2
- Participants With Phelan-McDermid Syndrome (PMS) at Week 4: Participants with Phelan-McDermid syndrome (PMS) at week 4
Arm/Group | Participants With Phelan-McDermid Syndrome (PMS) at Baseline | Participants With Phelan-McDermid Syndrome (PMS) at Week 1 | Participants With Phelan-McDermid Syndrome (PMS) at Week 2 | Participants With Phelan-McDermid Syndrome (PMS) at Week 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
seizure event | 22.6 (42.9) | 4.3 (7.8) | 15.8 (37.3) | 14.3 (33.2)

3. Secondary Outcome: Change in CGI - Improvement and Severity Scale
Description: Clinical Global Impressions (CGI) Rating Scales are commonly used to measure symptom severity and global improvement in treatment studies of patients with developmental disorders. There Severity Scale (CGI-S) is a 7-point scale (1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.) that requires the clinician to rate the severity of illness at the time of assessment. The Improvement Scale (CGI-I) is a 7-point scale (1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.) that requires the clinician to assess how much the illness has improved or worsened relative to baseline.
Time Frame: baseline, Week 1, Week 2, and Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Phelan-McDermid Syndrome (PMS) at Baseline | Participants With Phelan-McDermid Syndrome (PMS) at Week 1 | Participants With Phelan-McDermid Syndrome (PMS) at Week 2 | Participants With Phelan-McDermid Syndrome (PMS) at Week 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
score on a scale
  Improvement: number analyzed (Participants) | 06 | 6 | 6 | 6
  Improvement | 0 (0) | 0.83 (0.98) | 1 (1.1) | 1 (0.89)
  Severity | 5.33 (0.82) | 5.33 (0.82) | 5.33 (0.82) | 5.17 (0.75)

4. Secondary Outcome: Clinician-completed PMS Domain Specific Causes for Concerns Visual Analogue Scale (VAS)
Description: 9 item visual analogue scale completed by the clinician that scores the severity of concerns in domains that are clinically relevant in PMS. For each subject, the clinician is instructed to identify the top 4 or 5 that are of particular concern and that the clinician would most like to see change during the course of treatment with the study medication. The severity of the clinician's concern in each domain is scored by using a 10 cm visual analogue scale, with anchors of 0 "not at all severe" at the left and 100 "very severe" at the right end.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Phelan-McDermid Syndrome (PMS) at Baseline | Participants With Phelan-McDermid Syndrome (PMS) at Week 1 | Participants With Phelan-McDermid Syndrome (PMS) at Week 2 | Participants With Phelan-McDermid Syndrome (PMS) at Week 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
score on a scale
  Speech | 86.83 (8.13) | 84.33 (5.89) | 84.17 (5.85) | 81.67 (6.06)
  Thinking and Learning | 86.67 (6.83) | 77.5 (9.87) | 81.67 (6.83) | 78.33 (2.58)
  Seizures | 62 (28.43) | 41.67 (30.11) | 47.5 (34.31) | 44.17 (36.66)
  Gross Motor | 28.33 (28.23) | 26.67 (24.01) | 24.17 (22.45) | 25 (23.45)
  Repetitive Behavior | 70.33 (21.97) | 65 (24.08) | 60.83 (24.17) | 54 (25.77)
  Social Communication | 80.83 (8.61) | 77.5 (5.24) | 77.5 (6.89) | 74.17 (4.92)
  Sensory | 50.83 (21.78) | 48.33 (20.17) | 52.5 (22.97) | 50.33 (22.82)
  Activities of Daily Living | 78.33 (10.33) | 75 (10.95) | 76.5 (10.75) | 78.33 (8.76)
  Sleep | 43.33 (19.66) | 29.17 (17.15) | 43.33 (24.43) | 45 (30.66)

5. Secondary Outcome: Aberrant Behavior Checklist (ABC)
Description: rating scaled used to monitor an array of behavioral features among patients with intellectual disabilities. It takes 15-30 minutes to complete. 16 items, Each item is scored as 0 (never a problem), 1 (slight problem), 2 (moderately serious problem), or 3 (severe problem). with total from 0 to 48.
Time Frame: baseline, Week 1, Week 2, and Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Phelan-McDermid Syndrome (PMS) at Baseline | Participants With Phelan-McDermid Syndrome (PMS) at Week 1 | Participants With Phelan-McDermid Syndrome (PMS) at Week 2 | Participants With Phelan-McDermid Syndrome (PMS) at Week 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
score on a scale
  Irritability | 8.67 (6.02) | 9.33 (7.89) | 6.67 (3.72) | 4.83 (3.19)
  Lethargy | 15 (7.13) | 12 (7.9) | 9.83 (6.01) | 8.83 (4.96)
  Stereotypy | 6.67 (6.09) | 4.83 (5.08) | 4.17 (3.76) | 3.17 (2.93)
  Hyperactivity | 20.33 (11.34) | 14.33 (7.79) | 15.67 (9.09) | 13.83 (6.27)
  Inappropriate Speech | 1.17 (2.4) | 1.17 (2.4) | 0.17 (0.41) | 0 (0)

6. Secondary Outcome: Repetitive Behavior Scale-Revised (RBS-R)
Description: 42-item rating scale that is completed by a parent or caregiver. It reports on the severity of repetitive behaviors. each item scored on 4-point scale: 0-Behavior does not occur, 1-Behavior occurs and is a mild problem, 2-Behavior occurs and is a moderate problem, 3-Behavior occurs and is a severe problem. with total score from 0 (mild) to 126 (severe).
  Subscale ranges: stereotypic behavior (0 - 27);self-injurious behavior (0 - 24); compulsive behavior (0 - 18); ritualistic/Sameness Behavior (0 - 36); restricted Interests (0 - 9).
  Higher score in all subscales reflect increasing severity.
Time Frame: Baseline, Week 1, Week 2, Week 4
Population: Subjects received a single 6-hour intravenous infusion for a total dose administration or 120 mg/m2 of AMO-01.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Phelan-McDermid Syndrome (PMS) at Baseline | Participants With Phelan-McDermid Syndrome (PMS) at Week 1 | Participants With Phelan-McDermid Syndrome (PMS) at Week 2 | Participants With Phelan-McDermid Syndrome (PMS) at Week 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
score on a scale
  Stereotyped Behavior | 3.67 (3.5) | 3 (2.68) | 3.5 (2.07) | 2.67 (2.42)
  Self-Injury | 1.83 (1.94) | 1.33 (1.51) | 2 (2.45) | 1.5 (2.35)
  Compulsive Behavior | 2.5 (3.27) | 1.17 (1.47) | 2 (2.76) | 2.5 (2.81)
  Ritualistic Behavior | 0 (0) | 0.17 (0.41) | 0.17 (0.41) | 0 (0)
  Sameness Behavior | 2 (2.68) | 1.33 (1.75) | 2 (2.76) | 2.33 (2.66)
  Restricted Behavior | 1.83 (2.4) | 1.83 (2.04) | 1.67 (1.97) | 1.83 (2.56)
  Total | 11.83 (9.26) | 8.83 (5.56) | 11.33 (10.48) | 10.83 (10.87)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | AMO-01
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMO-01 (N=6)
Constipation (Gastrointestinal disorders) | 1
Sleep Issues (General disorders) | 1
Congestion/Cough (Respiratory, thoracic and mediastinal disorders) | 1
Headache (General disorders) | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Redness on hands (Skin and subcutaneous tissue disorders) | 1
Decreased appetite/weight loss (Metabolism and nutrition disorders) | 1
Viral Infection (Infections and infestations) | 1
Rash on nect (Skin and subcutaneous tissue disorders) | 1
Ear Infection (Ear and labyrinth disorders) | 1
Mouth movement, possible tic (Nervous system disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 2
Increased rubbing/repetitive behaviors (Psychiatric disorders) | 1
Seizure (Nervous system disorders) | 2
Drowsiness after infusion (Injury, poisoning and procedural complications) | 1
Flushing in face and hand (Injury, poisoning and procedural complications) | 1
Motor Stereotypes (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigators agree not to publish reports, abstracts, or other data compilations concerning the Study before the first multi-site publication by Sponsor. If there is no multi-site publication within 18 months after the Study has been completed or terminated at all Study locations, Principal Investigator shall have the right to publish and or present the results of the Study generated or collected at Study Site(s) (but not the results of any other Study location).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT03493607/Prot_SAP_000.pdf